CLINICAL TRIAL: NCT05420246
Title: The Efficacy and Safety of Ainuovirine in the Treatment of HIV-infected/AIDS Patients in China
Brief Title: Efficacy and Safety of Ainuovirine Treating With AIDS Patients
Acronym: ESATA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Linghua LI, Chief physician, Guangzhou 8th People's Hospital
Other Study IDs: X220314682
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: HIV/AIDS
Keywords: Ainuovirine Therapy;Real World Study;HIV-1-infected patients
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- These cases were given the treatment regimen including Ainuovirine: These cases were given the regimen including Ainuovirine (150mg, oral,qd)
  Interventions: Drug: Ainuovirine

INTERVENTIONS:
Drug: Ainuovirine — The regimen including Ainuovirine will be given to HIV-1 infected/AIDS patients.

SUMMARY:
Ainuovirine is the third generation of non nucleoside reverse transcriptase inhibitors(NNRTIs), for the treatment of HIV-1 infected adults. The existing clinical studies show that Ainuovirine is safe and potent, it solves the problem from the first-generation NNRTIs such as Efavirenz with large side effects and the second-generation like Rilpivirine not suitable for high viral load, but there are no relevant data or reports on the efficacy and safety of Ainuovirine in HIV-infected patients in China so far. This project aims to explore the efficacy and safety of ART regimens containing Ainuovirine for HIV-infected patients in real clinical environment, in further to guide clinical application.

DETAILED DESCRIPTION:
This study is an open-label, multicentered, single-arm and phase IV clinical trial.

450 HIV-infected patients who received Ainuovirine regimen (150mg, oral, qd) were included. At day 1 (1st collection as day 1), 3rd, 6th, 9th, 12th month, the rate of viral suppression and CD4+T cell count were calculated against baseline. In addition, the safety and drug compliance were also monitored.

Other indicators:

Demographic data (including gender, ethnicity, age, height, education level, occupation, route of infection), past medical history, smoking history, drug abuse history, hepatitis B markers, hepatitis C antibody, B ultrasound, chest X-ray, electrocardiogram, pregnancy test (Females of childbearing age): Day 1 (1st collection as Day 1), 1 time in total.

Vital signs (heart rate, blood pressure), body weight: 5 times on day 1 (the 1st collection was taken as day 1), 3rd, 6th, 9th, and 12th months.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of HIV infection 18-60 years old Patients who are prescribed to take Ainuovirine regimen . Sign informed consent

Exclusion Criteria:

1. Patients who are participating in other interventional clinical trials;
2. Patients who previously participated in the ACC007 study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who are prescribed to take including Ainuovirine regimen,because they are unable to tolerate the side-effect of or are not fit for the firstline free regimen in China,according to clinical judgment, no matter of the HIV-RNA viral loads and CD4 cell counts.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Virus suppression rate | 48 weeks
  ratio of HIV1-RNA < 20 copies/mL at 48 weeks of treatment
Adverse events | 48 weeks
  Any adverse events reported during the observational period

SECONDARY OUTCOMES:
Immune reconstitution indicators | 48 weeks
  CD4 cell count, CD4 +/ CD8 + ratio (baseline to 48 weeks)
Drug compliance | 48 weeks
  To explicit the number of people who have completed the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ruosu Ying, Doctor, Study Director — Guangzhou Eighth People's Hospital
Locations (1):
- Guangzhou 8th People's Hospital, Guangzhou Medical University., Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No